CLINICAL TRIAL: NCT06088121
Title: Effects of a ATNC MDD-V1 (TMS With Cognitive Training), for the Treatment of Mild Alzheimer Disease: a Randomized, Double-blinded, Placebo-controlled Study
Brief Title: Study to Evaluate the Efficacy and Safety of ATNC-MDD V1(TMS With Cognitive Training) in Mild Alzheimer's Dementia
Acronym: ATC-P001
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Advanced Technology & Communications (Industry)
Collaborators: Chungnam National University Hospital (Other); Korea University Anam Hospital (Other); Dong-A University Hospital (Other); Chonnam National University Hospital (Other); Chonbuk National University Hospital (Other); Chung-Ang University Gwangmyeong Hospital (Other); Yeungnam University Hospital (Other); Inje University Ilsan Paik Hospital (Other); National Health Insurance Service Ilsan Hospital (Other); Konkuk University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNUH 2023-03-027
Record Dates: First submitted 2023-09-19; First posted 2023-10-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer's Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorder
Keywords: TMS; Cognitive Stimulation; ATNC MDD-V1; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurodegenerative Diseases; Neurocognitive Disorders; Mental Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATNC MDD-V1 (Active Comparator): ATNC MDD-V1 treatment, synchronized TMS and cognitive training stimulation
  Interventions: Device: ATNC MDD-V1 (Real TMS + Real Cog); Device: ATNC BN-V1; Device: ATNC BN-V2
- Sham TMS + Real Cog (Sham Comparator): The Control arm subjects will receive daily treatments five days a week for 6 consecutive weeks of Sham treatment of TMS and real cognitive training which is similar to the real treatment in visit frequency and procedure.
  Interventions: Device: ATNC MDD-V1 (Sham TMS + Real Cog); Device: ATNC BN-V1; Device: ATNC BN-V2

INTERVENTIONS:
Device: ATNC MDD-V1 (Real TMS + Real Cog) — Synchronized TMS and cognitive stimulation to 6 brain areas.
  Other Names: ATNC MDD-V1; Brain Sense & Brain Cog
  Arms: ATNC MDD-V1
Device: ATNC MDD-V1 (Sham TMS + Real Cog) — Sham device, has the same appearance and sound as the real device, combined with real cognitive exercises. Patients come for the same number of sessions, delivers no real stimulation or cognitive training.
  Other Names: sham
  Arms: Sham TMS + Real Cog
Device: ATNC BN-V1 — The navigation system is used to determine the exact brain location to be stimulated (coordinates for the stimulation point).
  Other Names: Brain Navigation System V1
Device: ATNC BN-V2 — The navigation system is used to determine the exact brain location to be stimulated (coordinates for the stimulation point).
  Other Names: Brain Navigation System V2

SUMMARY:
The study tests the effect of the ATNC MDD-V1 on Alzheimer patients' cognitive function. The ATNC MDD-V1 uses non-invasive stimulation of both magnetic and cognitive training.

DETAILED DESCRIPTION:
The ATNC MDD-V1 system is a combined system of Transcranial Magnetic Stimulation and cognitive training and is a non-invasive therapeutic system for the improvement of Alzheimer patients' cognitive function.

A potential participant will undergo screening procedures to confirm eligibility to participate in the study, followed by randomization procedure to one of the study groups - treatment or sham (placebo) Patient will attend the clinic 5 times a week for 6 weeks, approximately an hour every day for treatment/sham. The patient will be required to return to the clinic for follow-up.

Up to 158 patients will be enrolled in up to 7 clinical sites in the Republic Korea.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who started drug treatment with an acetylcholinesterase inhibitor at least 2 months before participating in the clinical trial and can participate in the clinical trial without changing the dose during the trial period.
2. Male or female age 60-85 years.
3. Patients diagnosed with mild stage of Alzheimer's Disease, according to the NIA-AA (2011) diagnosis.
4. A patient whose dementia was confirmed to be due to Alzheimer's disease by amyloid PET-CT.
5. MMSE score 21 to 26.
6. CDR 1 or GDS 3.

   ※ For subjects who are excluded from screening based on criteria 5 or 6, if the investigator judges that the subject is likely to be eligible, one repeat screening may be performed.
7. A patient who is deemed physically eligible for the clinical trial based on medical records and physical examination.
8. A patient who is unable to provide voluntary informed consent for the clinical trial due to impaired decision-making capacity, for whom a legally authorized representative provides consent for participation, and who can attend follow-up visits with a caregiver.
9. Patients who agreed to participate in all 24-week clinical trials.
10. Patients with normal ability to see and hear letters.
11. Patients who speak Korean as their mother tongue

Exclusion Criteria:

1. Patients with central nervous system (CNS) disorders that may affect cognitive function (such as cerebrovascular diseases including vascular dementia, subdural hematoma, normal pressure hydrocephalus, brain tumors, CNS infections like HIV or syphilis, head trauma, Huntington's disease, Parkinson's disease, etc.) where cognitive decline may be explained by other causes, or in whom dementia types other than Alzheimer's disease are suspected.
2. Patients who have been unconscious due to brain surgery or concussion, or who have signs or symptoms of cranial pressure elevation on neurologic examination.
3. History of Epileptic Seizures or Epilepsy.
4. Patients with a history of drug abuse, including alcohol, in the past 5 years from the time of screening.
5. Patients with schizophrenia, schizoaffective disorder, bipolar disorder, current major depressive episode, psychosis, panic, post-traumatic stress, severe anxiety, mental retardation, DSM-V disorder.
6. Patients with abnormal vitamin B12, folic acid deficiency, or thyroid stimulating hormone (TSH) test results that were considered by the investigator to affect or are caused by the severity of dementia.
7. Patients with metal implants in the head, (i.e. cochlear implants, implanted brain stimulators and neurostimulators, aneurysm clips) with the exception of metal implants.
8. Cardiac pacemakers.
9. Implanted medication pumps.
10. Intracardiac lines.
11. Patients who are currently taking medications that lower the convulsive seizure threshold.
12. Significant heart disease.
13. Patients with severe renal or hepatic impairment※, referring to conditions that significantly affect daily living (e.g., stage 4 chronic kidney disease), with the assessment based on the investigator's judgment.
14. Contraindication for performing MRI scanning.
15. Contraindication for performing amyloid PET-CT scanning.
16. Patients who do not consent to TMS treatment and participation in this clinical trial.
17. Patients who participated in other clinical trials 3 months before participating in this clinical trial.

    ※ Subjects who participate in non-interventional studies (such as observational studies) that do not affect the subject's disease or symptoms may be enrolled in the study.
18. Patients with a history of TMS treatment within the last 2 years before participating in this clinical trial.
19. Patients judged by the investigator to be unsuitable for participation in clinical trials for other reasons.

    ※ If the test subject is unable to visit according to the research plan due to unavoidable personal circumstances during the screening period, it will be treated as a screening dropout, and the patient can participate in the study after re-agreeing according to the future schedule.
20. Patients with a history of malignant tumors within the last 5 years.

    - Participation is possible if more than 5 years have elapsed without recurrence after the decision to be cured (The point of complete removal of the tumor through surgery or the end of chemotherapy, etc.).
21. Patients who need to take medications suggested in concomitantly contraindicated drugs.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognition Score (Efficacy) | Week 24
  Change from Baseline to 24 weeks in ADAS-Cog score. ADAS-Cog: Alzheimer's Disease Assessment Scale - Cognitive

SECONDARY OUTCOMES:
Alzheimer's Disease Assessment Scale-Cognitive(ADAS-cog) Score (Efficacy) | Week 7, 12
  Change from Baseline to 7,12 weeks in ADAS-Cog score. ADAS-Cog: Alzheimer's Disease Assessment Scale - Cognitive
Korean-Mini Mental State Examination-2nd Edition(K-MMSE-2)(Efficacy) | Week 7, 12, 24
  Change from Baseline to 7, 12 and 24 weeks in K-MMSE-2. K-MMSE-2: Korean-Mini Mental State Examination-2nd Edition
Clinical Dementia Rating(CDR)(Efficacy) | Week 7, 12, 24
  Change from Baseline to 7, 12 and 24 weeks in CDR. CDR: Clinical Dementia Rating
Global Deterioration Scale(GDeps)(Efficacy) | Week 7, 12, 24
  Change from Baseline to 7, 12 and 24 weeks in GDeps. GDeps: Global Deterioration Scale
Clinical Global Impression of Change(CGIC)(Efficacy) | Week 7, 12, 24
  Change from Baseline to 7, 12 and 24 weeks in CGIC CGIC: Clinical Global Impression of Change
Korean-Instrumental Activities of Daily Living(K-IADL)(Efficacy) | Week 7, 12, 24
  Change from Baseline to 7, 12 and 24 weeks in K-IADL. K-IADL: Korean-Instrumental Activities of Daily Living

OTHER OUTCOMES:
Adverse events(AE's)(Safety) | Week 24
  Adverse events (AE's), including serious adverse events (SAEs) occurring at any time during the trial and follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ae Young MD LEE, PhD, Principal Investigator — Chungnam National University Hospital; Kun Woo MD Park, PhD, Principal Investigator — Korea University Anam Hospital; Deye MD Yoon, PhD, Principal Investigator — Dong-A University Hospital; Goun MD Kim, PhD, Principal Investigator — Chonbuk National University Hospital; Su-Hyun MD Jo, PhD, Principal Investigator — Chonnam National University Hospital; Mincheol MD Park, PhD, Principal Investigator — Chung-Ang University Gwangmyeong Hospital; Inwook MD Song, PhD, Principal Investigator — Incheon St.Mary's Hospital; Miyoung MD Park, PhD, Principal Investigator — Yeungnam University Hospital; Younggeon MD Lee, PhD, Principal Investigator — Inje University Ilsan Paik Hospital; Sohun MD Yoon, PhD, Principal Investigator — National Health Insurance Service Ilsan Hospital; Yeonsil MD Moon, PhD, Principal Investigator — Konkuk University Medical Center
Locations (11):
- South Korea (11):
  - Catholic university of Korea Incheon St. Mary's Hospital, Incheon, Bupyeong 6(yuk)-dong, Bupyeong-gu
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong, Deokan-ro 110
  - jeonbuk National University Hospital, Jeonju, Deokjin-gu
  - Chonnam National University Hopital, Gwangju, Dong-gu
  - Yeungnam University Medical Center, Daegu, Hyeonchung-ro, Nam-gu
  - National Health Insurance Service Ilsan Hospital, Gyeonggi-do, Ilsan-ro, Ilsandong-gu, Goyang-si
  - Inje University Ilsan Paik Hospital, Gyeonggi-do, Juhwa-ro, Ilsanseo-gu, Goyang-si
  - Chungnam National University Hospital, Daejeon, Jung-gu
  - Konkuk University Medical Center, Seoul, Neungdong-ro, Gwangjin-gu
  - Dong-A University Hospital, Busan, Seo-gu
  - Korea University Anam Hospital, Seoul, Seongbuk-gu

REFERENCES:
- See also: MedlinePlus Genetics related topics: Alzheimer disease — https://medlineplus.gov/genetics/condition/alzheimer-disease
- See also: MedlinePlus related topics: Alzheimer disease — https://medlineplus.gov/alzheimersdisease.html
- See also: Other U.S. FDA Resources — https://classic.clinicaltrials.gov/ct2/info/fdalinks
- See also: Sponsor's web — https://atnci.com